CLINICAL TRIAL: NCT06051149
Title: Effect of Catheter Type on Efficacy of Percutaneous Caudal Adhesolysis in Failed Back Surgery Syndrome.
Brief Title: Effect of Catheter Type on Efficacy of Percutaneous Caudal Adhesolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Abul-Fotouh Mohamed, principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUN1615
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Failed Back Surgery Syndrome
Keywords: caudal adhesiolysis; catheter type
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Intervention Model Description: double-blinded, prospective study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Will be performed in a sterile operating room under appropriate sterile precautions with help of assistant nurse who will open catheter set before principal investigator enter the operating room and the patient will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Epidural Catheter (Active Comparator): procedure Will be performed under sterile precautions utilizing fluoroscopy, RK needle.patient will be placed prone with a pillow under the abdomen.The sacral area draped from the top of the iliac crest to the bottom of the buttocks.The sacral Corns and the sacral hiatus will be palpated,is in the gluteal fold opposite the affected side will be infiltrated with lidocaine16gauge RK needle will be passed through the described entry point advanced to a point below the S3foramen to prevent S3nerve root damage.Placement will be confirmed by lateral and anteroposterior fluoroscopic views and after aspiration is negative for blood and CSF10mL of iohexol will be injected under fluoroscopy.Once the needle placement is confirmed to be in the epidural space, a lumbar epidurogram will be carried out utilizing approximately2to5 mL of contrast. then the bevel of the needle should face the ventrolateral aspect of the caudal canal.
  Interventions: Procedure: caudal adhesolysis using RACZ Catheter; Procedure: caudal adhesiolysis using NAVI Catheter
- RACZ Catheter (Active Comparator): same as procedure described above but using RACZ Catheter set
  Interventions: Procedure: caudal adhesolysis using RACZ Catheter
- NAVI catheter (Active Comparator): same as procedure described above but using NAVI Catheter set
  Interventions: Procedure: caudal adhesiolysis using NAVI Catheter

INTERVENTIONS:
Procedure: caudal adhesolysis using RACZ Catheter — caudal adhesolysis for patients with failed back surgery syndrome using RACZ Catheter under fluroscopy
  Arms: Epidural Catheter; RACZ Catheter
Procedure: caudal adhesiolysis using NAVI Catheter — caudal adhesolysis for patients with failed back surgery syndrome using NAVI Catheter under fluroscopy
  Arms: Epidural Catheter; NAVI catheter

SUMMARY:
The approach toward FBSS involves conservative management that consists of physical therapy and medication which aims to optimize gait and posture and can improve muscle strength and physical function

DETAILED DESCRIPTION:
The international association for the study of pain has defined failed back syndrome as persistent pain despite spine surgery in the same topographical area.

Several causes have been introduced for FBSS including pressure on the nerve root due to disc re-herniation or retained disc fragment, epidural fibrosis, acquired stenosis, and segmental instability.

Thus, FBSS is a syndrome with diverse etiologies and noticeable heterogeneity among patients. However, about 20% to 36% of FBSS occur due to epidural fibrosis, which is a progressive disease.

The approach toward FBSS involves conservative management that consists of physical therapy and medication which aims to optimize gait and posture and can improve muscle strength and physical function. Oral pharmacological treatment of FBSS is multimodal and increasingly controversial. Treatments include antiepileptics, non-steroidal anti-inflammatory drugs, oral steroids, antidepressants, and opioids including injections, and finally surgical options as a last line therapy. Other modalities including minimally invasive procedures like epidural injections, Epidural steroid injections (ESIs) are the most commonly performed procedure in pain clinics around the world. These can be administered primarily by three approaches: transforaminal, interlaminar, or caudally, and are indicated for symptoms of radiculopathy. Also radiofrequency ablation of nerves are often used to provide sustained relief that a diagnostic block or therapeutic injection cannot provide. Successfully targeting the intended nerve is achieved, maximizing the size of the lesion. Spinal cord stimulation (SCS) is a nother treatment modality that has shown tremendous potential in the management of FBSS. Adhesions can theoretically be lysed, thereby improving baseline pain scores and drug delivery of the ESI. Lysis of adhesions typically occurs by delivering hyaluronidase with hypertonic saline into the epidural space. The use of hyaluronidase with steroid may be more effective and have longer duration of effect than either one alone. Finally, surgical revision for FBSS is associated with a high morbidity with corresponding low rates of success.

Percutaneous adhesiolysis (PA), is a minimally invasive technique, that might be useful in the treatment of chronic pain refractory to conservative treatments. The basic idea behind PA is inserting a catheter in the ventral epidural space could directly break up perineural/epidural adhesions, that act as physical barriers to the perineurally deposited drugs but also cause neural irritation predisposing to neural inflammation.

ELIGIBILITY:
Inclusion Criteria:

* previous back surgery of at least 6 months duration.
* age ≥ 18.
* failure of conventional pharmacological management.

Exclusion Criteria:

* cauda equina syndrome.
* pregnant or lactating women.
* anti-coagulant therapy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
pain score | 6 months after intervention
  -difference in numeric rating scale at 6 months after intervention, minmal value 0 and maximum value 100 which is worst(more pain intensity)

SECONDARY OUTCOMES:
functional outcome | 6 months after intervention
  The Oswestry Disability Index,minmal value 0 and maximum value 50 which is worst(complete disability)

IPD SHARING:
Plan to Share IPD: No